CLINICAL TRIAL: NCT01448460
Title: Oocyte Vitrification for IVF Patients and Women With Fertility Threatening Conditions
Brief Title: Oocyte Vitrification for In Vitro Fertilization (IVF) Patients and Women With Fertility Threatening Conditions
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Greg L. Christensen, IVF Lab Director, University of Louisville
Other Study IDs: 09.356
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Fertility Preservation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: oocytes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fertility Patients: IVF patients with extra eggs or other subjects who desire egg vitrification for fertility preservation

SUMMARY:
Vitrification is a method of cryopreserving tissue for future use. It is widely used to preserve extra, good quality embryos generated from infertility treatments. It is becoming popular for the preservation of oocytes (eggs) as well, but is still considered investigational in this respect. The purpose of this study is to provide egg freezing for patients desiring fertility preservation. Although commonly used in clinics around the world, it should be offered as an IRB approved study procedure until it is no longer considered investigational by the American Society of Reproductive Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 37 and who require IVF for a successful pregnancy will be approached to consent for the study,. They must also have a cycle day 3 FSH < 10 mIU/ml, estradiol < 70 pg/ml and a baseline follicle count > 10. The BMI must be between 20 and 32kg/m2. If they do consent, eggs will only be vitrified if 13 or more mature metaphase II oocytes are collected.
* Women between the ages of 14 and 42 who are seeking treatment for fertility preservation. In addition they must also meet the following criteria.
* Patient is willing and able to delay any relevant therapy for up to 40 days.
* Have functioning ovaries as determined by blood / ultrasound testing.
* Patient is willing to undergo infectious disease testing for HIV, hepatitis B and C, syphilis, gonorrhea and Chlamydia.
* The patient must have clearance from their oncologist or medical specialist, if any, to undergo ovarian stimulation and transvaginal oocyte retrieval.
* The patient must not have a past history of blood clots in the veins or in the lungs.
* The patient must be willing to undergo transvaginal, internal ultrasound examination and pelvic examination.

Exclusion Criteria:

* Patients with a cycle day 3 FSH > 10 mIU/ml, cycle day 3 estradiol > 70 pg/ml and a baseline follicle count < 10 will be excluded.
* Patients with a BMI <20 and >32 will be excluded.
* Patients who are not willing or are unable to meet the above mentioned eligibility requirments.
* Patients with expected low ovarian reserve [evaluated on day 3 by an antral follicle count of <3 follicles at 2-5 mm diameter and/or an increased concentration of follicle stimulating hormone (FSH) >15 IU [15] on cycle day 3 ].
* Patients with possible poor quality of oocytes, based on medical history including previous exposure to chemotherapeutics or radiation.

Ages: 14 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: IVF patients who desire to have extra eggs, in excess of what is needed for their IVF cycle, or subjects requesting fertility preservation due to fertility threatening conditions such as cancer, advanced age or other.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)